CLINICAL TRIAL: NCT06437561
Title: Venous Aneurysm: a Case Series and Review of Literature
Brief Title: Report of Ten Cases of Venous Aneurysm in Extremities
Status: Completed | Type: Observational
Sponsor: Golestan University of Medical sciences (Other)
Responsible Party: Principal Investigator, Pezhman Kharazm, MD, Vascular Surgeon, Golestan University of Medical sciences
Other Study IDs: 114099
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Venous Aneurysm Nos; Arteriovenous Malformations; Vascular Diseases
Keywords: aneurysm; venous malformation; vascular surgery
MeSH Terms: conditions — Arteriovenous Malformations; Vascular Diseases; Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous aneurysms are not common in general, but because of the inherent risk of thrombosis in aneurysms, their timely diagnosis and treatment are recommended in most of the current sources. Ten cases of venous aneurysms were diagnosed and managed in our vascular surgery department from October 2018 to January 2024. Patient information was extracted from their files retrospectively.

DETAILED DESCRIPTION:
A vascular aneurysm is defined as the focal dilatation of a vessel. Aneurysm is classically used for arterial dilatations, although dilatations can occur in any part of the vascular system including veins. Venous aneurysms are not common in general, but with the increase in the use of duplex ultrasound, the number of cases diagnosed with venous aneurysms has recently increased. Venous aneurysms are more common in the lower limbs, and in the lower limbs, the involvement of the deep venous system is much more than the superficial venous system. According to reports, 77% of venous aneurysms are present in the lower limbs, of which 57% are in the deep venous system and 1.5% in the superficial venous system.

Considering their rarity, venous aneurysms may cause diagnostic challenges in some cases.

The importance of these aneurysms, especially in the lower limbs, which inherently have relative stasis due to the opposite flow direction of gravity, is that by creating venous stasis and whirlwind blood flow inside the aneurysm, they increase the susceptibility to clotting. Also, due to dysfunction of the pigeon nest valves, they cause chronic venous insufficiency. Although clot formation and subsequent pulmonary embolism are more common in deep venous aneurysms, cases of pulmonary embolism secondary to superficial venous aneurysms of the lower limbs have also been reported.

Complications caused by chronic venous insufficiency are more common in aneurysms that occur at the main junctions of superficial and deep veins, including saphenous femoral and saphenous popliteal junctions.

Considering the possible complications mentioned about venous aneurysms, these aneurysms need treatment, regardless of their location, and although in the superficial system, surgical resection is the most commonly recommended method, other surgical methods such as aneurysmectomy and primary repair, resection, and graft interposition, and also endovascular methods have been used. Of course, in case of insufficiency in the venous system, specific treatment of the cause of insufficiency (such as stripping of the large saphenous vein) is necessary in addition to the treatment of the aneurysm.

Regarding the follow-up after the treatment of aneurysms of the superficial system, most articles have recommended short-term treatment with anticoagulants and control of the superficial and deep systems through color doppler.

In this case series, we present 10 cases of venous aneurysms and discuss their presentation, diagnosis, and management.

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of venous aneurysm

Exclusion Criteria:

• Patient's non-consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with extremity venous aneurysm since 2018 to 2024
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
clinical presentation of extremity venous aneurysms | 6 years
  different clinical presentations of extremity venous aneurysms and their prevalence
age distribution of extremity venous aneurysms | 6 years
  prevalence of extremity venous aneurysms in different ages
location distribution of extremity venous aneurysms | 6 years
  prevalence of extremity venous aneurysms in upper vs. lower limbs as well as left side vs. right side
sex distribution of extremity venous aneurysms | 6 years
  prevalence of extremity venous aneurysms in both sexes

CONTACTS AND LOCATIONS:
Locations (1):
- Pezhman Kharazm, MD, Gorgan, Golestan Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code